CLINICAL TRIAL: NCT00965068
Title: Cholesterol in Autism Spectrum Disorder (ASD): Characterization and Treatment
Brief Title: Cholesterol in ASD: Characterization and Treatment
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 090203; 09-CH-0203
Record Dates: First submitted 2009-08-24; First posted 2009-08-25 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2015-06-08

CONDITIONS: Autism; Asperger Disorder; PDD-NOS
Keywords: Autism; Autism Spectrum Disorder; Cholesterol; Smith-Lemli-Opitz Syndrome; ASD; Pervasive Developmental Disorder; PPD-NOS
MeSH Terms: conditions — Autistic Disorder; Asperger Syndrome; Autism Spectrum Disorder; Smith-Lemli-Opitz Syndrome; Child Development Disorders, Pervasive | interventions — Cholesterol

INTERVENTIONS:
Other: Cholesterol

SUMMARY:
Background:

- Autism spectrum disorders (ASD) are developmental disabilities characterized by impaired social interaction and repetitive and/or stereotypical behaviors. Research studies suggest that some individuals with ASD have very low blood cholesterol levels. This low cholesterol level and other abnormal sterol levels may be important markers for

subtypes of ASD. Providing additional cholesterol to the diets of children with ASD may help improve behavior.

- These findings will guide the medical community in identifying individuals who should be tested for sterol disorders. This study will also help researchers learn whether adding extra cholesterol to the diet will improve behavioral and other autism spectrum characteristics seen in individuals with ASD and low cholesterol.

Objectives:

* To determine cholesterol levels in children with autism spectrum disorders.
* To compare behavioral and other characteristics among children who have autism spectrum disorders and high, low, or normal cholesterol levels.
* To determine whether adding cholesterol to the diet will improve behavioral and other characteristics in individuals with ASD and low cholesterol.

Eligibility:

- Children between the ages of 4 and 12 who have been diagnosed with an autism spectrum disorder.

Design:

* Initial screening study will involve a collection of blood samples (for study purposes and cholesterol testing).
* Children who have low cholesterol levels will take part in a study in which they will receive either cholesterol supplementation or a placebo, and will have detailed physical and psychological examinations to measure possible improvement in behavioral or other characteristics.
* Children who have high or normal cholesterol levels will have further blood samples taken, and will undergo an additional set of examinations for comparison purposes.
* Researchers may request blood or DNA samples from other family members (parents or siblings), which will be collected through blood draws and cheek swabs.

DETAILED DESCRIPTION:
Pilot work suggests that some individuals with autism spectrum disorders (ASD) have very low blood cholesterol levels. This low cholesterol level and other abnormal sterol levels may be important markers for subtypes of ASD. The proposed trial aims to characterize any clinical differences between low-cholesterol ASD and normal-or-high-cholesterol ASD and to test the response of individuals with ASD and low cholesterol to increased cholesterol in the diet.

Evidence for the role of low cholesterol in causing ASD in a subgroup of individuals comes from five sources. First, half of individuals with Smith-Lemli-Opitz syndrome (SLOS) meet the behavioral criteria for autistic disorder (Tierney et al, 2001), and three quarters have some type of ASD (Sikora et al, 2006). Second, in individuals with SLOS, the lower the cholesterol was in the blood and cerebrospinal fluid, the more severe were the autism and IQ and adaptive function deficits. Third, in SLOS, improvement was found in social and communication abilities with added dietary cholesterol. Fourth, cholesterol was low in a pilot study of 100 children with autism of unknown cause (Tierney et al, 2006). Fifth, it is becoming increasingly clear that cholesterol plays a pivotal role in several aspects of brain development.

This proposal is designed to 1) determine the prevalence of hypocholesterolemia in ASD individuals (ASD+Hypo); 2) determine the prevalence of hypercholesterolemia (in ASD individuals (ASD+Hyper); 3) determine the rate of SLOS in the ASD subjects; 4) determine the phenotype (physical, behavioral, and developmental) at less than the 5th centile (ASD+Hypo) and greater than the 95th centile (ASD+Hyper) individuals and normal cholesterol (ASD+Normal) in the ASD subjects; 5) test the efficacy of dietary cholesterol supplementation in ASD individuals with hypocholesterolemia; 6) determine whether a raised dose of cholesterol supplementation is more effective than a lower dose; and 7) create a repository of biomaterial samples from individuals with ASD and their biological family members.

Three sites (Kennedy Krieger Institute [KKI], Ohio State University [OSU], and the National Institutes of Health [NIH]) will collaborate to accomplish the objectives of this study. In addition to defining the frequency of altered cholesterol homeostasis in ASD, 60 youths (20 at each site) with ASD plus hypocholesterolemia will enter a 12-week, double-blind, placebo-controlled trial immediately followed by a 12-week open-label cholesterol trial to test the efficacy of dietary cholesterol supplementation. Outcome measures will include standard tests of behavior, communication, and other autism features.

These findings will guide the medical community in identifying individuals who should be tested for sterol disorders. This study will also help researchers learn whether adding extra cholesterol to the diet will improve behavioral and other autism spectrum characteristics seen in individuals with ASD and low cholesterol. The results of this study may help individuals with hypocholesterolemic ASD by the knowledge of the therapeutic value and safety of the use of cholesterol supplementation both biochemically and behaviorally. If improvement is demonstrated, it opens a new window to understanding the neurologic mechanisms of ASD. This knowledge may also be helpful for hypocholesterolemic individuals with ASD in that this newly identified population will benefit from such supplementation. Even if cholesterol supplementation is found to not be effective, important behavioral phenotype and developmental information will be obtained that might be useful in identifying subjects with ASD plus cholesterol abnormalities.

ELIGIBILITY:
* INCLUSION/EXCLUSION CRITERIA:

Screening Visit:

Inclusion:

* Parents agree to use a multivitamin with minerals if their child is selected to continue to the cholesterol supplementation clinical trial.
* Parents agree to not change the doses of other dietary supplement throughout the clinical trial, including megavitamins.
* Supplements or medications that are not meant to lower cholesterol levels but are likely to have cholesterol-lowering effects (such as Omega 3 or fish oil) will be permitted if the dose has been stable for at least 3 months prior to the initial screening visit.
* Male or female between the ages of 4.0-12.0 years at the time of consent/assent.
* Clinically diagnosed with an ASD for which no cause has been detected.
* Anticonvulsants used for the treatment of a seizure disorder will be permitted if the dosage has been stable for 3 months, and the subject is seizure free for at least 3 months.

Exclusion:

* Known pregnancy.
* Subject has SLOS or known cholesterol synthesis/regulation disorder.
* The subject has had an anticonvulsant dose change in the preceding 3 months or a seizure in the preceding 3 months.
* DSM-IV diagnosis of Rett Disorder, childhood disintegrative disorder, schizophrenia, another psychotic disorder, or substance abuse.
* A significant medical condition such as heart disease, hypertension, liver or renal failure, pulmonary disease, diabetes, or unstable seizure disorder identified by history, physical examination, or laboratory tests.
* Dietary supplementation doses, including megavitamins, have changed within the preceding 3 months.
* Currently on or has taken a statin or other medication meant to lower cholesterol within the preceding 3 months.
* Currently on or has taken dietary cholesterol supplementation within the preceding 3 months.
* Subjects will be excluded if they are on other medications or supplements that affect cholesterol or other lipid levels.
* Subjects with gastronomy feeding tubes (G-tubes) will be excluded.
* Subjects for whom English is not the primary language will be excluded.

(No subjects will be excluded based on race, ethnicity or gender).

Characterization Visit:

Inclusion:

* Same inclusion criteria as the Screening Visit.
* Participants must have a mental age of 18 months as measured at the Characterization Visit by the age-appropriate form of the Stanford Binet-V, the Differential Abilities Scale, or the Mullen Scales of Early Learning (N.B. potential subjects who test below 18 months of age, but are otherwise eligible, may be admitted to the study following a case review convened by the Multisite Steering Committee).
* Child must have an ASD diagnosis using DSM-IV and clinical judgment in order to proceed to the other components of the Characterization Visit.
* Neuroleptics will be permitted for the ASD+Hypo group only if the dosage remains stable for the duration of the study.
* Neuroleptic medication free for at least three months (ASD+Hyper and ASD+Normal only).

Exclusion:

* Same exclusion criteria as the Screening Visit.
* Allergy to lanolin or soy (Hypo+ASD only).
* Non-verbal mental age below 18 months as measured by the developmentally-appropriate form of the Stanford-Binet-V, Differential Abilities Scale, or the Mullen Scales of Early Learning (N.B. potential subjects who test below 18 months of age, but are otherwise eligible, may be admitted to the study following a case review convened by the Multisite Steering Committee).
* Did not meet the criteria for an ASD during the Characterization Visit.

Double-Blind, Placebo-Controlled trial phase for ASD+Hypo Only:

Inclusion:

* Met Characterization Visit inclusion criteria and completed Characterization Visit procedures.
* Met criteria for hypocholesterolemia in ASD.

Exclusion:

-Same exclusion criteria as the Characterization Visit.

Open-Label Trial for ASD+Hypo only:

Inclusion:

- Subject continues to meet double-blind, placebo-controlled trial phase inclusion criteria.

Exclusion:

- Subject started a neuroleptic medication or medication that affects cholesterol synthesis or metabolism.

Family Members of ASD+Hypo only:

Inclusion:

- Biological parent(s) and full or half-sibling(s) of any age.

Exclusion:

- Those individuals not willing to provide a blood sample or a saliva sample for DNA.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2009-07-28; Study Completion 2013-11-14 (Actual)

PRIMARY OUTCOMES:
Behavioral Changes

CONTACTS AND LOCATIONS:
Overall Officials: Forbes D Porter, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Irons M, Elias ER, Abuelo D, Bull MJ, Greene CL, Johnson VP, Keppen L, Schanen C, Tint GS, Salen G. Treatment of Smith-Lemli-Opitz syndrome: results of a multicenter trial. Am J Med Genet. 1997 Jan 31;68(3):311-4. PMID 9024565
- [Background] Elias ER, Irons MB, Hurley AD, Tint GS, Salen G. Clinical effects of cholesterol supplementation in six patients with the Smith-Lemli-Opitz syndrome (SLOS). Am J Med Genet. 1997 Jan 31;68(3):305-10. doi: 10.1002/(sici)1096-8628(19970131)68:33.0.co;2-x. PMID 9024564
- [Background] Kaufmann WE, Cortell R, Kau AS, Bukelis I, Tierney E, Gray RM, Cox C, Capone GT, Stanard P. Autism spectrum disorder in fragile X syndrome: communication, social interaction, and specific behaviors. Am J Med Genet A. 2004 Sep 1;129A(3):225-34. doi: 10.1002/ajmg.a.30229. PMID 15326621